CLINICAL TRIAL: NCT00912314
Title: A Randomized Trial of Maintenance Therapy With Posterior Tibial Nerve Stimulation for Overactive Bladder
Brief Title: Trial of Maintenance Therapy With Posterior Tibial Nerve Stimulation for Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0818191
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Overactive Bladder Syndrome
Keywords: OAB; overactive bladder; ptns; posterior tibial nerve stimulation; percutaneous tibial nerve stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive

ARMS (2):
- Monthly Maintenance PTNS (Active Comparator): After 12 weeks of PTNS, patients will be randomized to either the monthly PTNS arm, or the no maintenance PTNS arm.
  Interventions: Procedure: PTNS
- No maintenance PTNS (No Intervention): After 12 weeks of PTNS, patients will either be randomized to the Monthly PTNS arm or the No maintenance PTNS arm.

INTERVENTIONS:
Procedure: PTNS — Monthly PTNS after 12 weeks of weekly PTNS
  Arms: Monthly Maintenance PTNS

SUMMARY:
This study has 2 parts. Part 1 is a 12-week observational study of weekly Posterior Tibial Nerve Stimulation (PTNS) treatment for women with overactive bladder. Part 2 is a randomized, controlled trial of monthly maintenance PTNS therapy versus no therapy in subjects who were successfully treated by PTNS in Part 1.

Part 1: 12-week observational study of weekly PTNS treatment.

The primary aim of Part 1 is to determine the efficacy of a 12-week course of PTNS in the treatment of overactive bladder. Secondary aims are to determine the changes in voiding frequency and quality-of-life measures after the 12-week treatment.

Part 2: Randomized, controlled study of monthly PTNS compared to no PTNS after 12-week treatment

The primary aim is to determine time-to-failure after 12 weeks of PTNS in subjects who receive maintenance therapy compared to those who do not, in order to ascertain if there is a need for maintenance therapy after 12 weeks of PTNS. The investigators' secondary aims are to compare the long-term efficacy and quality of life impact in patient receiving maintenance PTNS compared to those that do not and to determine the efficacy of rescue maintenance PTNS in subjects who have symptom recurrence in the no maintenance therapy arm.

Hypothesis: There will be no difference in time to failure between women randomized to monthly maintenance PTNS compared to no maintenance PTNS.

DETAILED DESCRIPTION:
This study has two parts: an observational study of PTNS (Part 1) and a randomized, controlled trial of maintenance PTNS compared to no maintenance PTNS (Part 2).

Part 1: This is an observational study of the efficacy of PTNS therapy in women with bothersome OAB symptoms who have failed anticholinergic therapy. Subjects will be offered a standardized weekly regimen of PTNS for 12 weeks and asked to respond to surveys before and after treatment.

Pre- and post- intervention assessments will include a 3-day diary to assess voiding volume and frequency, Pelvic Floor Impact Questionnaire, Short Form Health Survey (SF-12), Patient Global Impression of Severity (PGI-S), Overactive Bladder Questionnaire (OAB-q short form bother),and the Pelvic Floor Distress Inventory Short Form (Urogenital Distress Inventory UDI 6 subset). Post-intervention assessment will include the above, as well as the Patient Global Impression of Improvement (PGI-I).

Part 2: After the initial 12-week treatment, all women with PGI-I less than 4, defined as patient perception of bladder function as better, much better, or very much better after the treatment than before the treatment, will be randomized to monthly PTNS or no PTNS. Part 2 of the study will continue for an additional 42 weeks (i.e. 52 weeks total in parts 1 and 2). Subjects will be considered to have failed therapy if their PGI-I score is greater than 3. If they are currently receiving PTNS maintenance therapy and have a PGI-I score greater than 3, they will be withdrawn from the study and transferred to clinical care to pursue other treatment options.

If they are in the no maintenance arm and have a PGI-I score greater than 3, then they are considered to have failed the no-maintenance treatment arm and may receive monthly PTNS treatment or pursue other treatment if they choose .

Study questionnaires will be administered to patients at clinic visits. PGI-I questionnaires will be administered via mail (followed by a phone call if the questionnaire is not received within a designated amount of time).

Sequence of Events

Part 1:

Initial urogynecology visit with history and physical (part of routine care). Identify patients interested in PTNS Offer participation in this study, at which point the subject visit transitions from routine care to a research visit.

Complete questionnaires and diaries to confirm inclusion criteria for those patients who opt to participate in this study.

Weekly PTNS sessions with nurse certified in PTNS administration for 12 weeks Telephone reminder to complete 3-day prospective voiding diary prior to MD visit.

In-person clinic visit with MD at end of 12-week treatment.

Part 2:

Clinic visit with MD at end of 12-week PTNS treatment, with administration of questionnaires. If PGI-I <4, then randomization to monthly maintenance or no maintenance.

Monthly RN visits for PTNS for those assigned to receive maintenance PTNS. Monthly administration of PGI-I by mail one week prior to scheduled PTNS treatment (or when it would be scheduled for those not randomized to receive it). If the questionnaire is not returned within one week, PGI-I will be administered by phone.

MD visit at one year for evaluation, administration of questionnaires, and end of study interview.

For patients who are already undergoing PTNS and therefore do not participate in Part 1 of the study, sequence of events will be as follows:

Clinic visit with MD at end of 12-week PTNS treatment. Identify patients interested in enrolling in the study. Offer participation and sign consents, at which point the subject visit transitions from routine care to a clinic visit.

Administration of questionnaires and voiding diary. If PGI-I <4, then randomization to monthly maintenance or no maintenance.

Monthly RN visits for PTNS for those assigned to receive maintenance PTNS. Monthly administration of PGI-I by mail one week prior to scheduled PTNS treatment (or when it would be scheduled for those not randomized to receive it). If the questionnaire is not returned within one week, PGI-I will be administered by phone.

MD visit at one year for evaluation, administration of questionnaires, and end of study interview.

PTNS Procedure:

In all study patients, PTNS will be performed per standard protocol by our trained clinical R.N. as follows. A 34-gauge needle is inserted approximately three fingerbreadths cephalad to the medial malleolus, between the posterior margin of the tibia and the anterior margin of the soleus muscle, approximately 3-4cm deep. A ground pad is applied on the same leg near the arch of the foot, and then the needle and electrode are connected to the Urgent PC stimulator (Urgent PC®, Uroplasty Inc., MN, USA), with an adjustable pulse intensity of 0-9 MA, a fixed pulse width of 200 microseconds, and a frequency of 20 Hz. The intensity is increased until the large toe starts to curl or the toes start to fan in order to assure correct placement, then turned down to an intensity the patient can tolerate. This treatment is performed in the clinic by a nurse trained in its administration, for 30 minutes weekly for 12 weeks. If the patient responds, then she is randomized to receive either 30-minute monthly maintenance treatment or no treatment.

Outcome Instruments

At baseline 12 weeks and 52 weeks,

3-day voiding diaries with frequency and volume charts

Questionnaires regarding quality of life and symptom improvement:

A. OAB-q (Overactive Bladder-q Short Form)

B. PFDI-SF (Pelvic Floor Distress Inventory Short Form)

C. PFIQ-SF (Pelvic Floor Impact Questionnaire Short Form)

D. PISQ-SF (Pelvic Organ Prolapse/Urinary Incontinence/Sexual Function Questionnaire Short Form)

E. SF-12 Medical Outcomes Study Short Form

F. PGI-I (Patient Global Impression of Improvement)

At week 12 and one week before their maintenance PTNS (or when their maintenance PTNS would be if they were randomized to receive it), patients fill out a mailed PGI-I.

Sample size

The primary outcome is time to failure as measured by PGI-I greater than 3. Because there is data for success rates with and without maintenance PTNS but no specific data regarding time to failure, we will use success rates to power the study. For 80% power, and a confidence level 0.05, if we estimate that 80% of people who initially respond to PTNS (as determined by PGI-I < 4) will continue to have improvement after 1 year with 12 weeks of PTNS followed by maintenance PTNS [Cooperberg 2005] and 20% will continue to have improvement for one year after 12 weeks of PTNS only [Nuhoglu 2006], then we need 7 subjects randomized to maintenance treatment and 7 subjects randomized to no maintenance treatment in Part 2. Based on the literature, we can expect at least 60% of subjects to respond to the 12-week course of PTNS, so we will need 23 subjects enrolled in Part 1 of the study. A sample size of 23 subjects at the start of Part 1 provides 14 responders for Part 2. This should offer 80% power to detect a relative difference of 50% between maintenance PTNS and no maintenance PTNS. To buffer against a potential drop-out rate over the year of 30%, we will plan to enroll 32 subjects total.

Secondary outcomes, including quality of life, condition-specific quality of life, and diary measures will be compared before and after the observational study, as well as at the end of the year. We will subcategorize subjects by whether or not they intended to remain on anticholinergic medications, whether or not they had detrusor overactivity based on urodynamic studies (if done), and whether those receiving PTNS after a year were originally randomized to receive maintenance PTNS or not.

Data management

At screening, each subject will be assigned a sequential study number. These will be de-identified and stored in locked file cabinets.

Block randomization will be performed in groups of 8 with a random number generator, and odd numbers assigned to PTNS maintenance, even numbers assigned to no maintenance PTNS. Assignments will be put in sequentially administered envelopes.

Statistical Analysis

The two groups will be compared with respect to demographic and baseline variables (e.g. age, race, BMI, quality of life status, prior treatment, current OAB medications) using chi squared and t tests.

Analysis of primary outcome will be a comparison of time to failure measured by PGI-I >3 in the group assigned to maintenance PTNS compared to the group not assigned to maintenance via chi-squared analysis. A cox regression model may be used to analyze time to failure on maintenance PTNS compared to no maintenance PTNS.

Other statistical and qualitative analyses will be performed on secondary outcome measures as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Women with refractory overactive bladder syndrome referred to UCSD Women's Pelvic Medicine Center by treating physician for PTNS therapy as standard of care
* At least 18 years old
* 9 or more voids per 24 hours
* PGI - S score of "moderate" or "great" bother
* If on anticholinergic medication, they must be on stable dose of medications for at least one month
* Able to provide informed consent and complete study measures

Exclusion Criteria:

* Postvoid residual > 150 ml to exclude subjects with urinary retention
* Active urinary tract infection (defer entry until resolved)
* Urine output > 2800 ml per day
* Diagnosis of interstitial cystitis or chronic pelvic pain
* Diagnosis of bladder cancer
* Currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
time-to-failure after 12 weeks of PTNS in subjects who receive maintenance therapy compared to those who do not | 40 weeks

SECONDARY OUTCOMES:
efficacy of a 12-week course of PTNS in the treatment of overactive bladder | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles Nager, MD, Principal Investigator — UCSD; Anna C Kirby, MD, Study Director — UCSD
Locations (1):
- UCSD Women's Pelvic Medicine Center, San Diego, California, United States